CLINICAL TRIAL: NCT05439486
Title: Evaluation the Efficacy and Safety of Hyperbaric Oxygen Therapy in Sildenafil Non Responder Erectile Dysfunction Patients.
Brief Title: New Treatment in Erectile Dysfunction Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Haisam Abdelrhman Ahmed Mohamed, Assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Soh-Med-22-01-38
Record Dates: First submitted 2022-05-20; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinded randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100% oxygen (Active Comparator): ED patients in this group exposed to hyperbaric oxygen 100 % concentration at 2.2 ATM for 90 minutes for 30 consecutive sessions.
  Interventions: Device: hyperbaric oxygen therapy within hyperbaric oxygen therapy chamber.
- ordinary room oxygen (Placebo Comparator): ED patients in this group exposed to normal air oxygen concentration at 2.2 ATM for 90 minutes for 30 consecutive sessions.
  Interventions: Device: hyperbaric oxygen therapy within hyperbaric oxygen therapy chamber.

INTERVENTIONS:
Device: hyperbaric oxygen therapy within hyperbaric oxygen therapy chamber. — ED patients in this group exposed to hyperbaric oxygen 100 % concentration at 2.2 ATM for 90 minutes for 30 consecutive sessions.

SUMMARY:
Erectile dysfunction patients who are non responder to sildenafil will be treated with hyperbaric oxygen therapy with 100% concentration and at 2 ATM for 30 consecutive sessions each one 90 minutes and then will be reassessed.

DETAILED DESCRIPTION:
This study is double blinded randomized controlled clinical trial that includes organic ED patients who attend to the Andrology out patient clinics, Department of Dermatology, Venerology and Andrology, Sohag University hospital, Sohag, Egypt. Informed consent was obtained from all patients. The study was submitted for approval by Ethical and Research committees at Sohag Faculty of Medicine, Sohag University, Sohag, Egypt.

Study design:

Patients were divided into two groups (randomly assigned and comparably cross matched for age). Both patients and the investigators were blinded as regard the treatment until the end of the study.

Group 1: Patients assigned to the HBOT group were treated with (30) sessions in consecutive days (90 minutes of 100% oxygen at 2.2 ATM).

Group 1: Patients assigned to control group were exposed to (30) sessions of air oxygen tension at 2.2 ATM.

All patients were subjected to the following:

1. Medical history:

   * Personal history: Age, residence, marital status, occupation and special habits of medical importance.
   * ED history: Onset, course and duration.
   * Sexual History: duration of marriage, wife age, frequency of intercourse, morning erection, orgasm, libido, percent of weakness, type and dose of PDE5I and its response after proper instructions and ejaculation.
   * Medical history : History of medical diseases (Hypertension, Diabetes mellitus, Liver disease and any chronic disease).
   * Therapeutic history: previous ED treatment modalities and response to them in addition to other current drug intake.
   * Past history of operations.
2. General examination:

   It included height, weight, BMI, Blood Pressure, hair distribution, fat distribution and breast examination.

   Blood pressure and pulse.
3. Local examination:

   Penis: (stretched flaccid length, urethral meatus, deformities and fibrosis). Testes: (site, size, consistency). Spermatic cord. Any scar of previous operations.
4. Erectile function evaluation:

   4-1- Arabic version of the sexual health inventory for men (SHIM): The SHIM is a five-item scale in which each item is scored from 0 to 5 on four items and 1 to 5 on one item. It includes four of the six items from the original erectile function domain of the IIEF and includes items in maintenance ability, erection confidence, maintenance frequency and erection firmness in addition to a single item on intercourse satisfaction.

   Among men in a relationship with a partner, including those men who have opportunity but no desire to attempt sexual activity or intercourse.

   Disease grades of ED on SHIM scores were categorized as follows: severe ED (SHIM score:1-7), moderate ED (8-11), mild-to-moderate ED(12-16), mild (17-21), and no ED (22-25). A cut off value of 21 was chosen, so that patients with scores of 21 or less were classified as having had ED while patients with scores above 21were classified as having no ED.

   4-2- Arabic version of Erection Hardness Score (EHS): The EHS is a single-item instrument that asks men to rate erection hardness on a scale that ranges from 0 (penis does not enlarge) to 4 (penis is completely hard and fully rigid).

   4-3- The sexual health encounter profile (SEP- Questions 2 and 3): The treatment efficacy evaluated through asking the patients to answer the SEP-Q2 and SEP-Q3 with yes or no.

   SEP-Q2: Were you able to insert your penis into your partner's vagina? SEP-Q3: Did your erection last long enough for you to have successful intercourse? 4-4- Penile color Doppler: Patients evaluated by penile color Doppler after intra-cavernosal injection of 1 ml of Prostaglandin E1 (10 µg/ml). Key parameters included PSV, (cavernosal artery blood flow rate at start of systole) and EDV, (cavernosal artery blood flow rate at the end of diastole.

   PSV <30 cm/s is considered evidence of arterial insufficiency (arteriogenic ED) and EDV >5 cm/s is consistent with venoocclusive ED.

   RI (defined as PSV-EDV/PSV) is an indicator for venoocclusive function assessment. RI >0.80 have been cited as indicative of normal veno-occlusive function.
5. Laboratory investigations:

   Patients evaluated with random blood sugar, lipid profile after 12 hours fasting, and serum uric acid. A morning 8:00- 10:00 a.m. blood sample collected for measurement of total and free testosterone.
6. Safety evaluation:

   Safety and tolerability evaluated throughout the course of the study by assessing adverse events reported by either the patient or the physician.
7. Follow up evaluation:

Patients evaluated at 3 points as follow:

The first initial evaluation, The second evaluation at the end of sessions and The third evaluation 3months after stoppage of sessions.

The evaluation tools were as follow:

Erectile function evaluation: SHIM- EHS- SEP- Penile color Doppler, Laboratory evaluation: Total and free testosterone and Safety evaluation.

Outcome measures:

The outcome measures were: SHIM- EHS- SEP- penile Doppler parameters - response to PDE5i- reported side effects by physician and /or patients.

Statistical analysis:

Data analyzed using Statistical Package for Social Sciences SPSS) software program (version 16). All variables checked for normality.

Quantitative variables with normal distribution presented as means ± standard deviation (SD). While quantitative variables with no normal distribution presented as median (25th-75th percentile). Qualitative variables recorded as frequencies and percentages .

Comparison between continuous variables with normal distribution done by student t- test, while continuous variables with no normal distribution done by Mann-Whitney test. Qualitative variables compared by chi-square test.

Correlations between different variable performed when indicated with appropriate tests. Regression analysis done if indicated.

P value < 0.05 considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with regular sexual relationship in the last 6 months
* having organic ED and
* non responder to Sildenafil were included in our study.

Exclusion Criteria:

* Hypogonadism,
* History of Pelvic trauma, surgery or disease,
* Receiving treatment in the last 3 months,
* History of premature ejaculation,
* History of spinal cord or brain disease,
* History of drug abuse,
* Patients without a regular sexual partner,
* Patients with advanced kidney disease (creatinine>1.3 mg\dl) or liver disease,
* History of psychiatric diseases,
* HBOT exclusion as open pneumo-thorax, chest disease, sezure and congestive heart failure.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-29 (Actual); Primary Completion 2022-08-29 (Estimated); Study Completion 2022-10-29 (Estimated)

PRIMARY OUTCOMES:
Change in sexual health inventory for men (SHIM) | Base line ( before the sessions), at the end of sessions (6 weeks after ) and then 3 months after.
  The SHIM is a five-item scale in which each item is scored from 0 to 5 on four items and 1 to 5 on one item. It includes four of the six items from the original erectile function domain of the IIEF and includes items in maintenance ability, erection confidence, maintenance frequency and erection firmness in addition to a single item on intercourse satisfaction.
  Among men in a relationship with a partner, including those men who have opportunity but no desire to attempt sexual activity or intercourse.
  Disease grades of ED on SHIM scores were categorized as follows: severe ED (SHIM score:1-7), moderate ED (8-11), mild-to-moderate ED(12-16), mild (17-21), and no ED (22-25). A cut off value of 21 was chosen, so that patients with scores of 21 or less were classified as having had ED while patients with scores above 21were classified as having no ED (Shamloul et al., 2004).
Change in Erection Hardness Score (EHS) | Base line ( before the sessions), at the end of sessions (6 weeks after ) and then 3 months after.
  The EHS is a single-item instrument that asks men to rate erection hardness on a scale that ranges from 0 (penis does not enlarge) to 4 (penis is completely hard and fully rigid) (Arafa and Shamloul, 2009).
Change in the Sexual health encounter profile (SEP- Questions 2 and 3): | Base line ( before the sessions), at the end of sessions (6 weeks after ) and then 3 months after.
  The treatment efficacy evaluated through asking the patients to answer the SEP-Q2 and SEP-Q3 with yes or no (Tsetsvadz A. et al., 2009).
  SEP-Q2: Were you able to insert your penis into your partner's vagina? SEP-Q3: Did your erection last long enough for you to have successful intercourse?

SECONDARY OUTCOMES:
Change in Penile color Doppler: | Base line ( before the sessions), at the end of sessions (6 weeks after ) and then 3 months after.
  Patients evaluated by penile color Doppler after intra-cavernosal injection of 1 ml of Prostaglandin E1 (10 µg/ml). Key parameters included PSV, (cavernosal artery blood flow rate at start of systole) and EDV, (cavernosal artery blood flow rate at the end of diastole) (Souper et al., 2017).
  PSV <30 cm/s is considered evidence of arterial insufficiency (arteriogenic ED) and EDV >5 cm/s is consistent with venoocclusive ED.
  RI (defined as PSV-EDV/PSV) is an indicator for venoocclusive function assessment. RI >0.80 have been cited as indicative of normal veno-occlusive function (Papagiannopoulos et al., 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Reham E Alsharkawy, Ass. prof., Study Chair — Sohag university- Faculty of Medicine; Amr A Ali, Ass. prof., Study Chair — Sohag university- Faculty of Medicine
Locations (1):
- Faculty of medicine sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No